CLINICAL TRIAL: NCT01866319
Title: A Multicenter, Randomized, Controlled, Three-Arm, Phase III Study to Evaluate the Safety and Efficacy of Two Dosing Schedules of Pembrolizumab (MK-3475) Compared to Ipilimumab in Patients With Advanced Melanoma
Brief Title: Study to Evaluate the Safety and Efficacy of Two Different Dosing Schedules of Pembrolizumab (MK-3475) Compared to Ipilimumab in Participants With Advanced Melanoma (MK-3475-006/KEYNOTE-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-006; 2012-004907-10 (EudraCT Number); MK-3475-006 (Other: Merck Protocol Number)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Melanoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ipilimumab (Experimental): Participants receive ipilimumab, 3 mg/kg intravenously (IV), once every 3 weeks (Q3W) for a total of 4 doses (up to approximately 3 months).
  Interventions: Biological: Ipilimumab
- Pembrolizumab Q2W (Experimental): Participants receive pembrolizumab, 10 mg/kg IV, once every 2 weeks (Q2W) for up to approximately 24 months.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab Q3W (Active Comparator): Participants receive pembrolizumab, 10 mg/kg IV, Q3W for up to approximately 24 months.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — 10 mg/kg IV, administered Q2W or Q3W based upon randomization.
  Other Names: MK-3475
  Arms: Pembrolizumab Q2W; Pembrolizumab Q3W
Biological: Ipilimumab — 3 mg/kg IV Q3W.
  Arms: Ipilimumab

SUMMARY:
This study will evaluate the safety and efficacy of 2 different dosing schedules of pembrolizumab (MK-3475), every 2 weeks (Q2W) and every 3 weeks (Q3W), and compare the 2 schedules to treatment with ipilimumab in ipilimumab-naïve participants with unresectable or metastatic melanoma. The primary hypotheses are that pembrolizumab is superior to ipilimumab with respect to progression-free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
Participants assigned to a primary course of pembrolizumab can receive up to 24 months of treatment. Participants with Stable Disease (SD) or better will then proceed to Post Treatment Follow-up. All efficacy and safety analyses will be based on the primary pembrolizumab course.

Participants who experience disease progression during the Post Treatment Follow-up will be eligible for a Second Course of pembrolizumab treatment for up to 1 additional year. With Amendment 05, all Second Course participants will be treated with a fixed dose of pembrolizumab 200 mg Q3W. With Amendment 06, after the study has achieved its key objectives or the study has ended, participants will be discontinued from this study and enrolled in an extension study to continue protocol-defined assessments and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of unresectable Stage III or metastatic melanoma not amenable to local therapy (excluding uveal or ocular melanoma)
* At least one measurable lesion
* No prior systemic treatment (excluding adjuvant or neoadjuvant therapy) for melanoma (first line) or one prior systemic treatment (excluding adjuvant or neoadjuvant therapy) for melanoma (second line)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Archived tissue sample or new biopsy sample
* Female participants of childbearing potential must agree to use effective contraception from Visit 1 to 120 days after the last dose of study drug; male participants must agree to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug

Exclusion criteria:

* Prior treatment with ipilimumab or other anti-cytotoxic T-Lymphocyte Antigen 4 (CTLA-4) agent or any anti-programmed cell death (PD-1 or PD-L2) agent
* Chemotherapy, radioactive, or biological cancer therapy within four weeks prior to the first dose of study drug, or not recovered from adverse events caused by cancer therapeutics administered more than four weeks earlier
* Currently participating or has participated in a study of an investigational agent or using an investigational device within 30 days of the first dose of study drug
* Expected to require any other form of systemic or localized antineoplastic therapy while on study
* On any systemic steroid therapy within one week before the planned date for first dose of randomized treatment or on any other form of immunosuppressive medication
* History of a malignancy (other than the disease under treatment in the study) within 5 years prior to first study drug administration, excluding adequately treated Stage 1 or Stage 2 basal/squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or other in situ cancers.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis; participants with previously treated brain metastases are eligible
* Severe hypersensitivity reaction to treatment with another monoclonal antibody
* Active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents
* Active infection requiring systemic therapy
* Known history of Human Immunodeficiency Virus (HIV)
* Known history of or positive for Hepatitis B or C
* Known psychiatric or substance abuse disorder
* Regular user (including recreational use) of illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)
* Pregnant or breastfeeding, or expecting to conceive, or father children within the projected duration of the study
* Received a live vaccine within 30 days prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2015-03-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Robert C,Schachter J,Long GV,Arance A,Grob JJ,Mortier L,Daud A,Carlino MS,McNeil C,Lotem M,Larkin J,Lorigan P,Neyns B,Blank CU,Hamid O,Mateus C,Shapira-Frommer R,Kosh M,Zhou H,Ibrahim N,Ebbinghaus S,Ribas A,KEYNOTE-006 investigators . Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Apr 19; PMID: 25891173
- [Result] Schachter J, Ribas A, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank C, Petrella TM, Hamid O, Zhou H, Ebbinghaus S, Ibrahim N, Robert C. Pembrolizumab versus ipilimumab for advanced melanoma: final overall survival results of a multicentre, randomised, open-label phase 3 study (KEYNOTE-006). Lancet. 2017 Oct 21;390(10105):1853-1862. doi: 10.1016/S0140-6736(17)31601-X. Epub 2017 Aug 16. PMID 28822576
- [Derived] Long GV, Carlino MS, McNeil C, Ribas A, Gaudy-Marqueste C, Schachter J, Nyakas M, Kee D, Petrella TM, Blaustein A, Lotem M, Arance AM, Daud AI, Hamid O, Larkin J, Yao L, Singh R, Lal R, Robert C. Pembrolizumab versus ipilimumab for advanced melanoma: 10-year follow-up of the phase III KEYNOTE-006 study. Ann Oncol. 2024 Dec;35(12):1191-1199. doi: 10.1016/j.annonc.2024.08.2330. Epub 2024 Sep 15. PMID 39306585
- [Derived] Robert C, Carlino MS, McNeil C, Ribas A, Grob JJ, Schachter J, Nyakas M, Kee D, Petrella TM, Blaustein A, Lotem M, Arance A, Daud AI, Hamid O, Larkin J, Anderson J, Krepler C, Grebennik D, Long GV. Seven-Year Follow-Up of the Phase III KEYNOTE-006 Study: Pembrolizumab Versus Ipilimumab in Advanced Melanoma. J Clin Oncol. 2023 Aug 20;41(24):3998-4003. doi: 10.1200/JCO.22.01599. Epub 2023 Jun 22. PMID 37348035
- [Derived] Hamid O, Robert C, Daud A, Carlino MS, Mitchell TC, Hersey P, Schachter J, Long GV, Hodi FS, Wolchok JD, Arance A, Grob JJ, Joshua AM, Weber JS, Mortier L, Jensen E, Diede SJ, Moreno BH, Ribas A. Long-term outcomes in patients with advanced melanoma who had initial stable disease with pembrolizumab in KEYNOTE-001 and KEYNOTE-006. Eur J Cancer. 2021 Nov;157:391-402. doi: 10.1016/j.ejca.2021.08.013. Epub 2021 Sep 25. PMID 34571336
- [Derived] Robert C, Hwu WJ, Hamid O, Ribas A, Weber JS, Daud AI, Hodi FS, Wolchok JD, Mitchell TC, Hersey P, Dronca R, Joseph RW, Boutros C, Min L, Long GV, Schachter J, Puzanov I, Dummer R, Lin J, Ibrahim N, Diede SJ, Carlino MS, Joshua AM. Long-term safety of pembrolizumab monotherapy and relationship with clinical outcome: A landmark analysis in patients with advanced melanoma. Eur J Cancer. 2021 Feb;144:182-191. doi: 10.1016/j.ejca.2020.11.010. Epub 2020 Dec 24. PMID 33360855
- [Derived] Lala M, Li TR, de Alwis DP, Sinha V, Mayawala K, Yamamoto N, Siu LL, Chartash E, Aboshady H, Jain L. A six-weekly dosing schedule for pembrolizumab in patients with cancer based on evaluation using modelling and simulation. Eur J Cancer. 2020 May;131:68-75. doi: 10.1016/j.ejca.2020.02.016. Epub 2020 Apr 15. PMID 32305010
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Robert C, Ribas A, Schachter J, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil CM, Lotem M, Larkin JMG, Lorigan P, Neyns B, Blank CU, Petrella TM, Hamid O, Su SC, Krepler C, Ibrahim N, Long GV. Pembrolizumab versus ipilimumab in advanced melanoma (KEYNOTE-006): post-hoc 5-year results from an open-label, multicentre, randomised, controlled, phase 3 study. Lancet Oncol. 2019 Sep;20(9):1239-1251. doi: 10.1016/S1470-2045(19)30388-2. Epub 2019 Jul 22. PMID 31345627
- [Derived] Wang M, Chen C, Jemielita T, Anderson J, Li XN, Hu C, Kang SP, Ibrahim N, Ebbinghaus S. Are tumor size changes predictive of survival for checkpoint blockade based immunotherapy in metastatic melanoma? J Immunother Cancer. 2019 Feb 8;7(1):39. doi: 10.1186/s40425-019-0513-4. PMID 30736858
- [Derived] Hamid O, Robert C, Ribas A, Hodi FS, Walpole E, Daud A, Arance AS, Brown E, Hoeller C, Mortier L, Schachter J, Long J, Ebbinghaus S, Ibrahim N, Butler M. Antitumour activity of pembrolizumab in advanced mucosal melanoma: a post-hoc analysis of KEYNOTE-001, 002, 006. Br J Cancer. 2018 Sep;119(6):670-674. doi: 10.1038/s41416-018-0207-6. Epub 2018 Sep 11. PMID 30202085
- [Derived] Carlino MS, Long GV, Schadendorf D, Robert C, Ribas A, Richtig E, Nyakas M, Caglevic C, Tarhini A, Blank C, Hoeller C, Bar-Sela G, Barrow C, Wolter P, Zhou H, Emancipator K, Jensen EH, Ebbinghaus S, Ibrahim N, Daud A. Outcomes by line of therapy and programmed death ligand 1 expression in patients with advanced melanoma treated with pembrolizumab or ipilimumab in KEYNOTE-006: A randomised clinical trial. Eur J Cancer. 2018 Sep;101:236-243. doi: 10.1016/j.ejca.2018.06.034. Epub 2018 Aug 7. PMID 30096704
- [Derived] Petrella TM, Robert C, Richtig E, Miller WH Jr, Masucci GV, Walpole E, Lebbe C, Steven N, Middleton MR, Hille D, Zhou W, Ibrahim N, Cebon J. Patient-reported outcomes in KEYNOTE-006, a randomised study of pembrolizumab versus ipilimumab in patients with advanced melanoma. Eur J Cancer. 2017 Nov;86:115-124. doi: 10.1016/j.ejca.2017.08.032. Epub 2017 Oct 4. PMID 28987768
- [Derived] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank CU, Hamid O, Mateus C, Shapira-Frommer R, Kosh M, Zhou H, Ibrahim N, Ebbinghaus S, Ribas A; KEYNOTE-006 investigators. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32. doi: 10.1056/NEJMoa1503093. Epub 2015 Apr 19. PMID 25891173
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=3475-006&kw=3475-006&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced melanoma were recruited to receive ipilimumab once every 3 weeks (Q3W), or a primary course of pembrolizumab administered every 2 weeks (Q2W) or every 3 weeks (Q3W).
Pre-assignment Details: 834 participants were randomized 1:1:1 to receive ipilimumab Q3W, pembrolizumab Q2W, or pembrolizumab Q3W. For participants receiving pembrolizumab, all safety and efficacy results data reported are for the primary pembrolizumab course received.
Groups:
- Ipilimumab: Participants received ipilimumab, 3 mg/kg intravenously (IV), once every 3 weeks (Q3W) for a total of 4 doses (up to approximately 3 months).
- Pembrolizumab Q2W: Participants received pembrolizumab, 10 mg/kg IV, once every 2 weeks (Q2W) for up to approximately 24 months.
- Pembrolizumab Q3W: Participants received pembrolizumab, 10 mg/kg IV, Q3W for up to approximately 24 months.
Period: Overall Study
Arm/Group | Ipilimumab | Pembrolizumab Q2W | Pembrolizumab Q3W
Started | 278 | 279 | 277
Treated | 256 | 278 | 277
Completed | 71 | 101 | 97
Not Completed | 207 | 178 | 180
Not completed — Adverse Event | 12 | 5 | 9
Not completed — Clinical progression | 3 | 2 | 2
Not completed — Death | 153 | 154 | 147
Not completed — Lost to Follow-up | 6 | 3 | 8
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 32 | 14 | 12

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population consisted of all randomized participants. Participants were included in the group to which they were randomized for Baseline Characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab | Pembrolizumab Q2W | Pembrolizumab Q3W | Total
Number analyzed (Participants) | 278 | 279 | 277 | 834
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (14.2) | 59.9 (14.6) | 61.2 (13.6) | 60.3 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 118 | 103 | 337
  Male | 162 | 161 | 174 | 497

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Independent Radiology Plus Oncology Review (IRO)
Description: PFS was defined as the time from randomization to the first documented disease progression, based on blinded Independent Radiology plus Oncology review (IRO) using RECIST 1.1, or death due to any cause, whichever occurred first. Disease progression was defined as a 20% or greater increase in the sum of diameters of target lesions with an absolute increase of at least 5 mm or the appearance of new lesions. The primary analysis of PFS was performed at the time of the first protocol pre-specified statistical analysis, with data cut-off of 03-Sep-2014.
Time Frame: Up to approximately 12 months (through first pre-specified statistical analysis cut-off date of 03-Sep-2014)
Population: The ITT population, comprising all participants as randomized to a study arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab | Pembrolizumab Q2W | Pembrolizumab Q3W
Number analyzed (Participants) | 278 | 279 | 277
Months | 2.8 [2.8 to 2.9] | 5.5 [3.4 to 6.9] | 4.1 [2.9 to 6.9]
Statistical Analysis 1: Comparison: Ipilimumab vs Pembrolizumab Q2W; Statistical testing was stratified by line of therapy (1st vs. 2nd), programmed cell death ligand 1 (PD-L1) status (positive vs. negative) and Eastern Cooperative Oncology Group (ECOG) performance status (0 vs. 1); Test type: Superiority or Other; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.46 to 0.72]
Statistical Analysis 2: Comparison: Ipilimumab vs Pembrolizumab Q3W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.47 to 0.72]
Statistical Analysis 3: Comparison: Pembrolizumab Q2W vs Pembrolizumab Q3W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.75869, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.21]

2. Primary Outcome: Percentage of Participants With Overall Survival (OS) at 12 Months
Description: OS was defined as the time from randomization to death due to any cause. The percentage of participants with OS (OS rate) at 12 months was reported for each arm. The reported percentage was estimated using a product-limit (Kaplan-Meier) method for censored data; data were censored at the date of cut-off. The primary analysis of OS was performed at the time of the second protocol pre-specified statistical analysis, with data cut-off of 03-Mar-2015.
Time Frame: Month 12
Population: The ITT population, comprising all participants as randomized to a study arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab | Pembrolizumab Q2W | Pembrolizumab Q3W
Number analyzed (Participants) | 278 | 279 | 277
Percentage of participants | 58.2 [51.8 to 64.0] | 74.1 [68.5 to 78.9] | 68.4 [62.5 to 73.6]
Statistical Analysis 1: Comparison: Ipilimumab vs Pembrolizumab Q2W; Statistical testing was stratified by line of therapy (1st vs. 2nd), PD-L1) status (positive vs. negative) and ECOG performance status (0 vs. 1); Test type: Superiority or Other; p = 0.00052, Regression, Cox; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.47 to 0.83]
Statistical Analysis 2: Comparison: Ipilimumab vs Pembrolizumab Q3W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.00358, Regression, Cox; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.52 to 0.90]
Statistical Analysis 3: Comparison: Pembrolizumab Q2W vs Pembrolizumab Q3W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.51319, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI [0.67 to 1.22]

3. Secondary Outcome: Objective Response Rate (ORR) According to RECIST 1.1 as Assessed by IRO
Description: ORR was defined as the percentage of the participants with a best tumor response of complete response (CR: disappearance of all target lesions with any pathological lymph nodes having a reduction in short axis to <10 mm) or partial response (PR: ≥30% decrease in the sum of diameters of target lesions), based on IRO using RECIST 1.1. The primary analysis of ORR was performed at the time of the first protocol pre-specified statistical analysis, with data cut-off of 03-Sep-2014.
Time Frame: Up to approximately 12 months (through first pre-specified statistical analysis cut-off date of 03-Sep-2014)
Population: The ITT population, comprising all participants as randomized to a study arm.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ipilimumab | Pembrolizumab Q2W | Pembrolizumab Q3W
Number analyzed (Participants) | 278 | 279 | 277
Percentage of Participants | 11.9 [8.3 to 16.3] | 33.7 [28.2 to 39.6] | 32.9 [27.4 to 38.7]
Statistical Analysis 1: Comparison: Ipilimumab vs Pembrolizumab Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.00013, Miettinen & Nurmimen; Percent difference = 16.1, 95% CI 2-sided [7.8 to 24.5]
Statistical Analysis 2: Comparison: Ipilimumab vs Pembrolizumab Q3W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.00002, Miettinen & Nurmimen; Percent difference = 17.2, 95% CI 2-sided [9.5 to 25.6]
Statistical Analysis 3: Comparison: Pembrolizumab Q2W vs Pembrolizumab Q3W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.82636, Miettinen & Nurmimen; Percent difference = -1.1, 95% CI [-10.6 to 8.6]

ADVERSE EVENTS:
Time Frame: Up to approximately 69 months (through End of Trial Analysis data cut-off date of 03-Jun-2019)
Description: All-Cause Mortality table includes all randomized participants.
  Serious and Other adverse events (AEs) tables include all randomized participants who received at least 1 dose of study drug. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Ipilimumab | Pembrolizumab Q2W | Pembrolizumab Q3W
All-Cause Mortality (participants affected / at risk) | 173/278 | 166/279 | 162/277
Serious Adverse Events (participants affected / at risk) | 77/256 | 89/278 | 90/277
Other Adverse Events (participants affected / at risk) | 220/256 | 257/278 | 247/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab (N=256) | Pembrolizumab Q2W (N=278) | Pembrolizumab Q3W (N=277)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Anaemia aggravated (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Lymph nodes enlarged (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Decompensation cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Heart attack (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Paroxysmal atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0)
Adrenomegaly (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Panhypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Neovascular glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blood in stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 16 (18) | 6 (6) | 6 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 7 (7) | 3 (3)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage of digestive tract (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis aggravated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Partial small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sigmoiditis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anasarca (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue aggravated (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 4 (4) | 1 (1) | 0 (0)
General body pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 1 (1)
Reduced general condition (General disorders) | 1 (1) | 0 (0) | 0 (0)
Unknown cause of death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 4 (4) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Cellulitis aggravated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis of oral soft tissues (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis of upper arm (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Central line infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Meningoencephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Myelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septicaemia gram-negative NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Shoulder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound breakdown (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Bilirubin total increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hyponatremia aggravated (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain aggravated (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hips osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in heel (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pathologic fracture of femur (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pathologic fracture of humerus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Prolapsed lumbar disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Unilateral leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
B-cell chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (7) | 2 (2)
Basal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Desmoplastic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Epidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Huerthle cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intra-epidermal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intracranial tumour bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Signet-ring cell adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Superficial basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid papillary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsions aggravated (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage brain (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Horner's syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraneoplastic limbic encephalitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression aggravated (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute renal insufficiency (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (2)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bullous lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bullous pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Drug rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Poor venous access (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis leg (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vein disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab (N=256) | Pembrolizumab Q2W (N=278) | Pembrolizumab Q3W (N=277)
Anaemia (Blood and lymphatic system disorders) | 12 (14) | 34 (44) | 23 (28)
Hyperthyroidism (Endocrine disorders) | 6 (6) | 17 (19) | 12 (12)
Hypothyroidism (Endocrine disorders) | 5 (5) | 29 (31) | 25 (26)
Abdominal pain (Gastrointestinal disorders) | 16 (19) | 29 (37) | 18 (19)
Constipation (Gastrointestinal disorders) | 29 (32) | 53 (78) | 39 (47)
Diarrhoea (Gastrointestinal disorders) | 69 (91) | 82 (162) | 76 (116)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 26 (27) | 20 (21)
Nausea (Gastrointestinal disorders) | 55 (66) | 73 (90) | 70 (88)
Vomiting (Gastrointestinal disorders) | 31 (35) | 45 (66) | 27 (32)
Asthenia (General disorders) | 26 (29) | 45 (92) | 41 (56)
Fatigue (General disorders) | 73 (78) | 90 (125) | 85 (116)
Fever (General disorders) | 20 (22) | 29 (40) | 21 (35)
Flu-like symptoms (General disorders) | 8 (9) | 21 (23) | 14 (27)
Common cold syndrome (Infections and infestations) | 9 (9) | 21 (32) | 15 (18)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 31 (43) | 21 (25)
Urinary tract infection (Infections and infestations) | 10 (11) | 22 (33) | 14 (19)
Alanine aminotransferase increased (Investigations) | 12 (13) | 21 (32) | 16 (19)
Aspartate aminotransferase increased (Investigations) | 12 (13) | 22 (35) | 12 (17)
Lactate dehydrogenase increased (Investigations) | 6 (6) | 14 (25) | 6 (11)
Weight decreased (Investigations) | 13 (13) | 20 (21) | 26 (28)
Anorexia (Metabolism and nutrition disorders) | 24 (27) | 31 (39) | 35 (36)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 16 (34) | 13 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (18) | 41 (63) | 39 (42)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 29 (32) | 11 (12)
Knee pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 15 (21) | 8 (8)
Low back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 17 (19) | 12 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 32 (38) | 15 (18)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 21 (26) | 12 (12)
Dizziness (Nervous system disorders) | 9 (9) | 27 (34) | 22 (26)
Headache (Nervous system disorders) | 27 (29) | 45 (72) | 33 (58)
Anxiety (Psychiatric disorders) | 4 (4) | 14 (14) | 10 (10)
Insomnia (Psychiatric disorders) | 14 (14) | 28 (33) | 20 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 58 (75) | 43 (48)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (10) | 15 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 30 (32) | 27 (27)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 16 (16) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 19 (20) | 17 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 65 (76) | 68 (99) | 59 (83)
Rash (Skin and subcutaneous tissue disorders) | 28 (29) | 37 (55) | 36 (51)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (8) | 17 (23) | 10 (15)
Vitiligo (Skin and subcutaneous tissue disorders) | 4 (4) | 34 (36) | 42 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.